CLINICAL TRIAL: NCT05869370
Title: The Effects Of Low Intensity Training With Blood Flow Restriction In The Lower And Upper Limbs On Muscle Strength, Muscle Mass, Biochemical Parameters And Markers Of Systemic Inflammation In Rheumatoid Arthritis Patients: A Randomized Clinical Trial
Brief Title: The Effects Of Low Intensity Training With Blood Flow Restriction In Rheumatoid Arthritis Patients
Acronym: TBFR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital de Clínicas de Porto Alegre (Unknown)
Responsible Party: Principal Investigator, Ricardo Machado Xavier, PhD, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0071
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Kaatsu; Blood Flow Restriction Training
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity resistance training (Experimental)
  Interventions: Other: High intensity resistance training
- Low intensity resistance training combined with blood flow restriction (Experimental)
  Interventions: Other: Low intensity resistance training combined with blood flow restriction

INTERVENTIONS:
Other: High intensity resistance training — Twelve weeks of resistance training twice a week.
  Arms: High intensity resistance training
Other: Low intensity resistance training combined with blood flow restriction — Twelve weeks of resistance training with blood flow restriction twice a week.
  Arms: Low intensity resistance training combined with blood flow restriction

SUMMARY:
Rheumatoid arthritis (RA) patients showed systemic manifestations that may lead to a reduction in muscle strength, muscle mass and, consequently, to a reduction in physical function. On the other hand, high intensity resistance training (HIRT) are able to improve muscle strength and muscle mass in RA without affecting the disease course. However, due to the articular manifestations caused by this disease, these patients may present intolerance to HIRT. Thus, the low intensity resistance training with blood flow restriction (TBFR) may be a new training strategy for these populations. In this sense, the investigators speculate that TBFR could be beneficial in RA patients, as well as, HIRT.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Rheumatoid arthritis patients;
* All individuals will undergo an ergospirometry to ensure cardiorespiratory conditions.

Exclusion Criteria:

* Fibromyalgia;
* Cardiovascular disease;

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-05-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | Twelve weeks
  1 maximum repetition test.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio Grande do Sul - Faculdade de Medicina - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Dos Santos LP, Santo RCDE, Ramis TR, Portes JKS, Chakr RMDS, Xavier RM. The effects of resistance training with blood flow restriction on muscle strength, muscle hypertrophy and functionality in patients with osteoarthritis and rheumatoid arthritis: A systematic review with meta-analysis. PLoS One. 2021 Nov 10;16(11):e0259574. doi: 10.1371/journal.pone.0259574. eCollection 2021. PMID 34758045